CLINICAL TRIAL: NCT03428451
Title: Prophylaxis Versus Treatment Against TURP Syndrome : Role of Hypertonic Saline
Brief Title: Prophylaxis Versus Treatment for TURP Syndrome.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ahmed Mohamed ELbadawy (Other)
Responsible Party: Sponsor-Investigator, Ahmed Mohamed ELbadawy, Ahmed Mohamed ELbadawy- Clinical investigator , Cairo University, Kasr El Aini Hospital
Organization: Kasr El Aini Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N02112
Record Dates: First submitted 2018-01-26; First posted 2018-02-09 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Transurethral Resection of Prostate Syndrome
Keywords: TURP; hypertonic saline; TURP syndrome; hyponatraemia
MeSH Terms: conditions — Hyponatremia | interventions — Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Hypertonic saline ) (Active Comparator): patients will receive NaCl 3% HS at a dose of 4 ml/kg/hr.
  Interventions: Drug: NaCl 3% HS
- Group B (Hypertonic saline) (Active Comparator): patients will receive NaCl 3% HS at a dose of 2 ml/kg/hr.
  Interventions: Drug: NaCl 3% HS
- Group C (Normal saline) (Active Comparator): patients will receive NaCl 0.9% NS at a dose of 6 ml/kg/hr.
  Interventions: Drug: NaCl 0.9% NS

INTERVENTIONS:
Drug: NaCl 3% HS — Hypertonic saline 3% is a type of crystalloid solution with osmolarity higher than that of plasma.
  Other Names: Hypertonic saline
  Arms: Group A (Hypertonic saline )
Drug: NaCl 3% HS — Hypertonic saline 3% is a type of crystalloid solutions with osmolarity higher than that of plasma.
  Other Names: Hypertonic saline
  Arms: Group B (Hypertonic saline)
Drug: NaCl 0.9% NS — Normal saline 0.9% is a type of crystalloid solution with osmolarity similar to that of plasma.
  Other Names: Normal saline
  Arms: Group C (Normal saline)

SUMMARY:
This study is designed to investigate the usage & effects of prophylactic HS preloading, with two different concentrations, to combat the expected dilutional hyponatremia induced by irrigating fluid absorption and to prevent the occurrence of TURP syndrome with its potential complications

DETAILED DESCRIPTION:
The study will be conducted on 60 patients ASA class I - III BPH patients, candidates for TURP surgery using monopolar electronic resectoscope. Eligible patients will be allocated into one of three study groups (n=20 in each). Group A patients will receive NaCl 3% HS at a dose of 4 ml/kg/hr; Group B patients will receive NaCl 3% HS at a dose of 2 ml/kg/hr; while Group C patients will receive NaCl 0.9% Normal Saline(NS) at a dose of 6 ml/kg/hr. All intra-venous infusions will be started 30 minutes before the subarachnoid block, and continued all through the procedure at the same specific rate for each infusion. Vital signs [mean BP, HR, CVP & oxygen saturation (spO2)] will be recorded. Plasma electrolytes (sodium, potassium, chloride)and serum osmolality (mOsm) will be measured. Incidence of TUR syndrome, need for ICU admission, post-operative ventilation and total hospital stay will be noted.

ELIGIBILITY:
Inclusion Criteria:

* ASA class I - III BPH patients

Exclusion Criteria:

* Patients having any condition contra-indicating regional anesthesia e.g impaired coagulation.
* Electrolyte imbalance,
* Uncontrolled hypertension,
* Congestive heart failure or being allergic to local anesthetics.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Adult male BPH patients
Enrollment: 60 (Estimated)
Dates: Start 2018-02-10 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Serum sodium level measured in mEq/L | 72 hours
  Hyponatremia was defined as a serum sodium < 130 mEq/L

SECONDARY OUTCOMES:
Incidence of TURP syndrome | 72 hours
  Occurring TURP syndrome manifestations
Need for ICU admission | 72 hours
  For cardio-pulmonary support(vasopressor,mechanical ventilation), neurological monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed ELbadawy, MD, Principal Investigator — Faculty of medicine- Cairo University- Egypt
Locations (1):
- Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided